CLINICAL TRIAL: NCT01222871
Title: Treatment of Early Nasal Polyposis With Topical Triamcinolone
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: not enough particpants
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Peter Catalano, Chief of Otolaryngology, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00540
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Nasal Polyps
Keywords: Treatment
MeSH Terms: conditions — Nasal Polyps | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 study groups, experimental and control.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triamcinolone (Experimental): Triamcinolone soaked nasopore dressing
  Interventions: Drug: Triamcinolone
- Control Group (Placebo Comparator): Saline soaked sponge
  Interventions: Drug: Saline soaked sponge

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone soaked nasopore dressing
  Other Names: Kenalog (40)
  Arms: Triamcinolone
Drug: Saline soaked sponge — saline soaked sponge
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare the effectiveness of intranasal Triamcinolone delivered through a bio-absorbable nasal dressing verses oral steroids and a saline soaked dressing, in the treatment and prevention of early nasal polyposis.

DETAILED DESCRIPTION:
nasopore, a bio-absorbable nasal dressing, may offer an alternative route of sustained steroid drug delivery. The use of topical targeted intranasal steroids may prevent the routine adverse effects of oral steroids while maintaining the same therapeutic / clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with early nasal polyposis

Exclusion Criteria:

* Age < 18 years
* Patients with active sinus infections
* Patients on long term steroids
* Allergy or sensitivity to steroids
* Patients with Antrochoanal polyps
* Patients who received topical steroids by bio-resorbable sponge or oral steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Catalano, MD, Study Director — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- St. Elizabeth's Medical Center, 736 Cambridge St, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject enrolled but study was terminated and subject did not start the study.
Groups:
- Triamcinolone: Nasopore Triamcinolone soaked sponge
- Control: Saline soaked sponge
Period: Overall Study
Arm/Group | Triamcinolone | Control
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone | Control | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — No participant started because study was terminated.
Sex: Female, Male — No participant started because study was terminated.

OUTCOME MEASURES:

1. Primary Outcome: Nasal Endoscopic Exam Findings .
Description: nasal endoscopic exam findings at 2 weeks, 6 weeks and 12 weeks were not collected from any participant.
Time Frame: 2 weeks, 6 weeks, 12 weeks were not collected from any participant.
Population: No participant started because study was terminated.
Arm/Group | Triamcinolone | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: no data collected, Study terminated.
Description: No data collected, study terminated.
Groups:
- Saline Soaked Sponge: Nasopore saline soaked sponge
Arm/Group | Triamcinolone | Saline Soaked Sponge | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No